CLINICAL TRIAL: NCT03618238
Title: A Pilot Study of Anlotinib for the Evaluation of Safety and Efficacy in Patients With Stage IV Natural Killer/T-cell Lymphoma and Refractory to L-asparaginase Based Chemotherapy
Brief Title: Anlotinib for Advanced and Refractory Natural Killer /T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Rong Tao, Clinical Professor and Associate Director of Department of Hematology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHLSG-NK-1604
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type
Keywords: anlotinib; L-asparaginase resistant
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Intervention Model Description: drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental): patients will be given anlotinib 12 mg daily for continus 14 days every 21 days until disease progression.
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — 12 mg daily for continus 14 days every 21 days
  Other Names: Anlotinib Hydrochloride

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of anlotinib in patients with stage IV extranodal natural killer/T-cell lymphoma, nasal type.

DETAILED DESCRIPTION:
Extranodal natural killer/T-cell lymphoma (ENKTCL), nasal type, is a rare subtype of non-Hodgkin lymphoma (NHL) with relatively high incidence in China. L-asparaginase based chemotherapy improved overall response and prolonged the long-term survival for patients with stage IV. But the treatment for the patients with advanced disease and resistant to L-asparaginase based chemotherapy has not been established. The overall survival for these patients are very poor. This study is designed to evaluate the efficacy and safety of anlotinib in patients with stage IV ENKTCL and refractory to L-asparaginase based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of extranodal natural killer/T-cell lymphoma, nasal type.
* stage IV disease and resistant to L-asparaginase-based combined chemotherapy.(Definition of L-asparaginase resistance: Progression during treatment or no response to treatment).
* Eastern Cooperative Oncology Group (ECOG ) performance status 0~3.
* Preserved organ functions for: absolute neutrophil counter (ANC)>1.0×109/L, Platelet>50×109/L, hemoglobin>80g/L, total bilirubin (TBIL)<2×ULN, alanine transaminase (ALT)<2×ULN, normal serum creatinine，fibrinogen≥1.0g/L, LVEF≥50%.
* Signed Informed consented.

Exclusion Criteria:

* patients with a disease resistant to L-asparaginase but may benefit from a radiotherapy.
* HIV, hepatitis virus C (HCV), or active hepatitis virus B (HBV) infection with HBV DNA≥105 copies/ml.
* Significant complications: autoimmune disease, severe infection, or liver cirrhosis, hemophagocytic lymphohistiocytosis, disseminated intravascular coagulation, uncontrolled hypertension or diabetes, hemorrhagic or thrombotic events within 6 months.
* Mental disorders.
* Pregnant or lactation
* Peptic ulcer
* Enrolled in other trial treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 12 weeks after the initiation of anlotinib treatment
  The treatment response will be assessed every 12 weeks.

SECONDARY OUTCOMES:
Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Day 1 of each course and then every 3 months for 2 years
  Treatment-Related Adverse Events will be assessed and graded by NCI CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No